CLINICAL TRIAL: NCT02479789
Title: Efficacy of Intravenous Lidocaine in the Operative Management of Thyroid Surgery With Intraoperative Nerve Monitoring
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bronx-Lebanon Hospital Center Health Care System (Other)
Responsible Party: Principal Investigator, Ramasamy Govindarajan, Clinical Research In-Charge, Anesthesia, Bronx-Lebanon Hospital Center Health Care System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 04091501
Record Dates: First submitted 2015-06-21; First posted 2015-06-24 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Thyroidectomy; Nerve Monitoring
Keywords: Intravenous Lidocaine; Recurrent laryngeal nerve; Intra operative nerve monitoring; Thyroidectomy
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Experimental): Subjects in the Lidocaine arm of the randomized trial will receive a bolus of 1 mg /Kg of IV lidocaine followed by 1.5 mg/KG/h of IV lidocaine infusion during the surgery which will be stopped at extubation.
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Subjects in the Placebo arm of the randomized trial will receive a bolus of 1mg/kg Placebo ( 0.9% saline) followed by 1.5 mg/KG/h Placebo ( 0.9% saline) infusion during the surgery which will be stopped at extubation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine
  Other Names: Xylocaine, Lignocaine
  Arms: Lidocaine
Drug: Placebo
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
Intra operative Nerve Monitoring ( IONM ) is rapidly becoming the standard of care for thyroid surgery to prevent injury to the recurrent laryngeal nerve. However the laryngo tracheal reflexes need to be adequately suppressed to permit proper utilization of intra operative nerve monitoring. Increasing the depth of anesthesia to achieve this often leads to side effects. Intravenous lidocaine infusion has been shown to be effective in blunting these reflexes. The planned study intends to look at the efficacy of intravenous lidocaine infusion in decreasing the amount of anesthesia medications needed to suppress the reflexes. Also the study looks at the analgesic and anti emetic properties of intravenous lidocaine infusion post operatively by measuring these outcomes.

The study is designed as a double blinded randomized controlled trial with 30 subjects in the group who will receive intravenous lidocaine during surgery and 30 subjects in the group who will receive placebo. Blunting of the laryngo tracheal reflexes intra operatively will be recorded as the primary outcome. The amount of anesthesia medications, the post operative patient comfort level, pain control, usage of narcotic pain medications, nausea, vomiting will be recorded as secondary outcomes.

DETAILED DESCRIPTION:
Intra Operative Nerve Monitoring ( IONM) is rapidly becoming a standard of care in many institutions across the country. While the overall incidence of nerve palsy is low, when it occurs it is a devastating lifelong handicap . Several studies have documented that routine identification of the RLN with IONM has decreased the rates of permanent RLN palsy It is not designed to visualize the recurrent laryngeal nerve (RLN), but to allow intra-operative assessment of RLN function as well as to establish a prognosis in patients developing RLN paralysis. Complete functionality of the IONM depends on near total laryngeal relaxation and reflex suppression without the use of neuromuscular blocking agents (NMBAs). The depth of anesthesia required to meet that criteria often leads to hemodynamic instability.

When the IONM signal is unchanged after the resection, the surgeon can be reassured that postoperative vocal cord function is normal in 99.6% of cases. Where the IONM signal is absent or abnormal, 30-45% of the patients will develop vocal cord dysfunction postoperatively The successful deployment and data analysis from the IONM depends upon the complete laryngeal relaxation and reflex suppression. The IONM causes strong contractions of the vocal cords and is an independent cause of laryngeal alterations . The surgical procedure is a strong factor of stress to the larynx with a potentially traumatic manipulation at the level of the larynx . Complete functionality of the IONM constitutes before the full electromyographic recovery of the NMB at the adductor pollicis muscle , as the laryngeal muscles recover faster than the peripheral muscles . The anesthetic technique chosen should ensure absolute laryngeal reflex suppression as the effect of the short acting depolarizing muscle relaxant is wearing off immediately following intubation, until preferably the extubation. Be it total intravenous anesthesia or inhalation-based anesthesia, the depth required for reflex suppression can cause profound cardiovascular instability. While the attempts to titrate down the anesthetic depth can cause resurfacing of the troublesome laryngeal reflexes, attempts to counter the side effects with sympathomimetic agents can themselves result in a myriad of undesirable hemodynamic consequences. The resulting hemodynamic fluctuations can result in adverse outcomes in patients with significant cardiovascular co-morbidities.

Laryngoscopy with or without intubation, provokes a sympathoadrenal response. These events are especially detrimental in individuals who have limited myocardial reserve because of age or disease; these include geriatric population and those with significant coronary arteriosclerosis as in diabetes mellitus, sustained hypertension, angina, ischemic heart disease and cardiac dysrhythmias . IV lidocaine decreases the intracellular Ca2+ concentration in airway smooth muscle, decreases myofilament Ca2+ sensitivity and has been shown to suppress coughing and prevent reflex broncho constriction. Injected intravenously, lidocaine is variably effective in blunting the hemodynamic response to tracheal intubation .

IV lidocaine has analgesic, anti-hyperalgesic and anti-inflammatory properties. Local anesthetics can reduce the postoperative inflammatory response in several ways such as blocking neural transmission at the site of tissue injury and thus attenuating neurogenic inflammation. In addition because of anti-inflammatory properties of their own, they may inhibit the migration of granulocytes and release of lysosomal enzymes, consequently leading to a decreased release of pro-inflammatory cytokines. Pro-inflammatory cytokines can induce peripheral and central sensitization, leading to pain augmentation (hyperalgesia)

Because of its plasma half life of 8 min, an IV bolus of 1 - 1.5 mg/kg lidocaine must be followed by infusion of 1 - 4 mg/min in adults in order to maintain therapeutic levels of 1.5 - 4 μg/mL (15, 16). Lidocaine side effects have never been reported in its intended use, probably because the first clinical signs of toxicity occur at considerably high blood concentrations (> 5 μg/mL), which did not occur even when IV lidocaine was given continuously over 14 days . Lidocaine infusion at the rate of 1.5 mg/kg/h following a bolus of 1.5 mg/kg has been employed in a newborn to perform an intra-operative wake-up test during neurosurgery . It was also used during thyroidectomy in 60 y old patient with cardiac co morbidities This will be a prospective double blinded randomized controlled trial done at Bronx Lebanon Hospital Center. 60 consecutive patients undergoing thyroidectomy using nerve monitoring will be randomized into two groups of thirty each. One group will receive IV Lidocaine infusion during the surgery to facilitate the nerve monitoring. The other group will receive a placebo.

Patient recruitment:

The nurse administrator in the General Surgery clinic will talk to all patients coming to the clinic for thyroid surgery and will inform them about the study. A booklet explaining the nature of the study, risks and benefits will be provided to the patients by the administrator. Patients who are willing to participate in the study will be asked to convey the same with the surgeon.

After this the patients will be sent for pre operative medical evaluation and testing. Based on the history, physical examination, investigations and medical evaluation, they will be included or excluded from the study.

Informed consent will then be taken from the patients willing to participate in the study and those who meet the inclusion criteria. This consent will be separate from the surgical consent.

The day of surgery:

The patient will come to ambulatory surgery after overnight fasting. Vitals will be checked and the patient is seen by the anesthesiologist and surgeon in the ambulatory surgery unit. There after the patient is wheeled into the operating room for surgery.

Two days prior to the surgery, pharmacy will be notified of the case. The research pharmacist will prepare the lidocaine or placebo vial according to the randomization chart. This will be picked up and given to the anesthesiologist.

In the operating room:

The surgery is done in supine position with the head extended using a shoulder roll. Propofol and Fentanyl are used for induction. Neuro muscular blockade which is routinely used in other surgeries will not be used in this surgery.

Dragonfly Single Channel Laryngeal Surface Electrode (Electrode LSE 500Ms; Neurovision Medical Products,Ventura, CA, USA) will be applied to a #7 cuffed ETT (Medline Industries, Mundelein, Illinois, USA) according to the manufacturer's instructions. The patient will be pre-oxygenated and then induced with a bolus of midazolam 2 mg and fentanyl 1.25 μg/kg followed by etomidate 0.25 mg/kg and succinylcholine 1.2 mg/kg intravenously. Direct laryngoscopy is done and endotracheal intubation is done. The nerve monitoring apparatus is set up and the placement of the electrode plates touching the vocal cords will be verified under vision with a Glidescope®, after positioning the patient with the desired neck extension or by impedence measurement. The patient will be cleaned and draped.The patients will receive a bolus of 1 mg /Kg of IV lidocaine/Placebo ( 0.9% saline) followed by 1.5 mg/KG/h of IV lidocaine/Placebo ( 0.9% saline) infusion during the surgery which will be stopped at extubation.

Esmolol in titrated boluses will be used to blunt the sympatho adrenal responses during the intubation. Anesthesia will be maintained with 50:50 mixture of air in oxygen and 1 - 2 minimum alveolar concentration of sevoflurane. IV infusion of propofol 50 μg/ kg/min will be titrated to effect for maintenance. Intra operative nerve monitoring ( IONM) will be used to identify the recurrenct laryngeal nerves. Dragonfly Single Channel Laryngeal Surface Electrode [Neurovision Medical Products, Ventura, CA; Electrode LSE 500Ms] will be used as part of the electromyography circuit to facilitate the neve monitoring. A Bispectral Index (BIS) monitor (Aspect Medical Systems, Newton, MA; Model 1 A 2000) will be used to guard against "recall" during lighter planes of anesthesia and a train of four (TOF) monitor [ Microstim Plus, Neurotechnology, Houston, Texas, USA ] will be employed to guard against inadvertent neuromuscular blockade.

The study is designed as a double blinded randomized controlled trial with 30 subjects in the group who will receive intravenous lidocaine during surgery and 30 subjects in the group who will receive placebo. The intended period of the study will be one year. Blunting of the laryngo tracheal reflexes intra operatively will be recorded as the primary outcome. The amount of anesthesia medications, the post operative patient comfort level, pain control, usage of narcotic pain medications, nausea, vomiting will be recorded as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients undergoing bilateral thyroid surgery
* Age- 18-85 y

Exclusion Criteria:

* Patients undergoing additional procedures,
* Patients younger than 18y or older than 85 years.
* Patients at high risk for use of lidocaine due to Congestive heart failure, arrhythmia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-06; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Suppression of laryngo tracheal reflexes during thyroid surgery | From beginning of surgery to the end of surgery
  Number of times laryngo tracheal reflexes were encountered during surgery will be recorded.

SECONDARY OUTCOMES:
Amount of Anesthesia medications used | From beginning of surgery to the end of surgery
  The total amount of each anesthesia medication used will be recorded
Post operative pain control | At 30 minutes, two hours, eight hours, 24 hours after surgery
  Pain will be measured on a scale of 1 to 10
Post operative usage of medications to control pain | Within 24 hours of surgery
  The total amount of medications used to control pain will be recorded
Post operative nausea | At 30 minutes, two hours, eight hours, 24 hours after surgery
  Number of episodes of nausea and vomiting will be recorded
Post operative overall patient comfort as measure of the anti inflammatory effect of Lidocaine | At 30 minutes, two hours, eight hours, 24 hours after surgery
  Comfort level will be measured on a scale of 1 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Ramasamy Govindarajan, MD, Principal Investigator — Bronx Lebanon Hospital Center
Locations (1):
- Health and Wellness Center- Bronx Lebanon Hospital Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Study still recruiting

REFERENCES:
- [Result] Govindarajan R, Shah A, Reddy VS, Parithivel V, Ravikumar S, Livingstone D. Improving the functionality of intra-operative nerve monitoring during thyroid surgery: is lidocaine an option? J Clin Med Res. 2015 Apr;7(4):282-5. doi: 10.14740/jocmr2025w. Epub 2015 Feb 9. PMID 25699129